CLINICAL TRIAL: NCT02856204
Title: Shotgun Sequencing for Etiologic Diagnosis of Febrile Neutropenia
Brief Title: Shotgun Sequencing in Diagnosing Febrile Neutropenia in Patients With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: HEMAML0035; NCI-2016-01128 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 32817 (Other: Stanford IRB)
Record Dates: First submitted 2016-08-02; First posted 2016-08-04 (Estimated); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Acute Myeloid Leukemia; Febrile Neutropenia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Febrile Neutropenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples

GROUPS / COHORTS (1):
- Diagnostic (collection of blood samples): Patients undergo collection of blood samples before and during the episode of febrile neutropenia for up to 6 weeks.
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Cytology Specimen Collection Procedure — Undergo collection of blood
  Other Names: Cytologic Sampling
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This research trial studies the shotgun sequencing of blood samples in diagnosing febrile neutropenia in patients with acute myeloid leukemia. Studying samples of blood from patients with acute myeloid leukemia in the laboratory may help identify pathogens and accurately diagnose infections such as febrile neutropenia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test the hypothesis that shotgun metagenomics is not inferior to standard of care diagnostics in the detection of pathogens in patients with febrile neutropenia.

SECONDARY OBJECTIVES:

I. To establish a microbiological diagnosis with known or unknown pathogens in patients in whom standard care failed to yield a pathogenic diagnosis.

OUTLINE:

Patients undergo collection of blood samples before and during the episode of febrile neutropenia for up to 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with febrile neutropenia
* A primary diagnosis of acute myeloid leukemia (AML)

Exclusion Criteria:

* Prior history of febrile neutropenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospitalized patients (at Stanford Hospital and Clinics) with acute myelogenous leukemia (AML), who are expected to have neutropenia (defined as absolute neutrophil count < 500 / cubic mm) lasting ≥ 7 days after chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2016-08; Primary Completion 2017-12 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Detection of pathogens in patients with febrile neutropenia assessed by shotgun metagenomics | Up to 6 weeks
  Will be compared to standard of care diagnostics in the detection of pathogens in patients with febrile neutropenia.
Number and frequency of novel pathogens found | Up to 6 weeks
Proportion of patients with any pathogen by the standard, where the shotgun did not indicate the presence of the pathogen | Up to 6 weeks
Proportion of patients with false negative | Up to 6 weeks
Proportion of patients with false positives | Up to 6 weeks
Proportion of patients with mitochondrial DNA detected | Up to 6 weeks

SECONDARY OUTCOMES:
Microbiological diagnosis with known or unknown pathogens in patients in whom standard care failed to yield a pathogenic diagnosis assessed by shotgun metagenomics | Up to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Deresinski, Principal Investigator — Stanford University; Steven Coutre, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Palo Alto, California, United States